CLINICAL TRIAL: NCT02324153
Title: A Randomized Double Blind Placebo Controlled Trial of Ramelteon in the Prevention of Post-operative Delirium in Older Patients Undergoing Orthopedic Surgery
Brief Title: Ramelteon in the Prevention of Post-operative Delirium
Acronym: RECOVER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00097232; 1R21AG050850-01A1 (NIH)
Record Dates: First submitted 2014-12-15; First posted 2014-12-24 (Estimated); Results first posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Delirium; Delirium, Dementia, Amnestic, Cognitive Disorders; Delayed Emergence From Anesthesia; Cognitive Disorders
Keywords: Post-operative Delirium
MeSH Terms: conditions — Delirium; Neurocognitive Disorders; Delayed Emergence from Anesthesia; Cognitive Dysfunction; Emergence Delirium | interventions — ramelteon; microcrystalline cellulose; Riboflavin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Ramelteon 8 mg oral dose Riboflavin 100 mg (preoperative first dose only)
  Interventions: Drug: Ramelteon; Drug: Microcrystalline Cellulose; Drug: Riboflavin 100 mg
- Placebo (Placebo Comparator): Capsule Shells filled with microcrystalline cellulose Riboflavin 100 mg (preoperative first dose only - if received as an outpatient)
  Interventions: Drug: Microcrystalline Cellulose; Drug: Riboflavin 100 mg

INTERVENTIONS:
Drug: Ramelteon — 1 pre-operative and 2 nightly postoperative doses of Ramelteon/placebo will be administered
  Other Names: Rozerem
  Arms: Treatment
Drug: Microcrystalline Cellulose — Placebo Comparator
Drug: Riboflavin 100 mg — Riboflavin will be added to both placebo and active intervention capsules in order to track adherence to dose while taken as an outpatient (i.e. only the first preoperative dose)
  Other Names: Adherence marker

SUMMARY:
This trial focuses on a Phase II randomized masked clinical trial testing the effectiveness and safety of peri-operative administration of ramelteon, a melatonin agonist in the prevention of postoperative delirium.

DETAILED DESCRIPTION:
This trial will randomize older aged patients undergoing general or regional anesthesia for orthopedic surgical procedures to three perioperative doses of a melatonin agonist, ramelteon, and placebo in a masked double blind fashion. The primary outcomes are 1) the incidence of post-operative delirium in the recovery period in the Postoperative Anesthesia Care Unit and on post-operative days 1 and 2 following surgery, and 2) the safety of ramelteon as documented by the presence of adverse events in the follow-up period.

ELIGIBILITY:
* Planned orthopedic surgery under general or regional anesthesia and post-operative inpatient stay
* 65 years of age or older
* Mini-mental Status Exam (MMSE) score of 15 or greater prior to surgery;
* Ability to understand, speak, read and write English.

Exclusion Criteria:

* Delirium diagnosis on the Confusion Assessment Method instrument at baseline
* Is unable to give informed consent due to cognitive impairment and a suitable legally authorized representative (LAR) cannot be identified
* Declines participation
* Current medications that include:

  1. ramelteon
  2. melatonin
  3. fluvoxamine
  4. rifampin
  5. ketoconazole
  6. fluconazole
* History of ramelteon or riboflavin intolerance
* Heavy daily alcohol intake by medical record or history
* Current moderate to severe liver failure (as defined by Charlson criteria
* Evidence of Systemic Inflammatory Response Syndrome (SIRS) as measured by > 2 criteria8)
* Presence of a condition that in the opinion of the PI compromises patient safety or data quality if enrolled in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin J Neufeld, MD MPH, Principal Investigator — Professor - Department of Psychiatry and Behavioral Sciences
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh ES, Leoutsakos JM, Rosenberg PB, Pletnikova AM, Khanuja HS, Sterling RS, Oni JK, Sieber FE, Fedarko NS, Akhlaghi N, Neufeld KJ. Effects of Ramelteon on the Prevention of Postoperative Delirium in Older Patients Undergoing Orthopedic Surgery: The RECOVER Randomized Controlled Trial. Am J Geriatr Psychiatry. 2021 Jan;29(1):90-100. doi: 10.1016/j.jagp.2020.05.006. Epub 2020 May 16. PMID 32532654

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 41 | 39
Completed | 33 | 38
Not Completed | 8 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Surgery postponed after randomization | 3 | 0
Not completed — Developed delirium preoperatively | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients randomized to either treatment with ramelteon or placebo
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 33 | 38 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.3 (5.5) | 75.4 (5.0) | 74.9 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 14 | 14 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 27 | 32 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 38 | 71
DRS-R98 Total [Mean (Standard Deviation); unit: units on a scale] — Delirium Rating Scale-Revised-98(23) Severity items are rated on a scale of 0-3 and diagnostic items are rated on a scale of 0-2 or 0-3. The minimum score is 0. The maximum possible score for severity items is 39, while the maximum total score is 46. Higher scores indicate more severe delirium; score of 0 indicates no delirium.
  units on a scale | 2.2 (2.6) | 2.6 (3.0) | 2.4 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Delirium During Two Days Following Surgery
Description: Delirium DSM 5 based criteria informed by standardized history gathering, examination, cognitive evaluation using cognitive tests, informant interview, and medical record review) measured during Post-operative Day 1 and/or Day 2
Time Frame: Up to Post Operative Day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 33 | 38
Participants | 3 | 2

2. Primary Outcome: Number of Participants With Delirium in the Post Anesthesia Care Unit (PACU)
Description: Delirium (DSM 5 based criteria informed by standardized history gathering, examination, cognitive evaluation using cognitive tests, informant interview, and medical record review) measured once recovered from anesthesia.
Time Frame: Post Operative Day 0: Post Anesthesia Care Unit Following Recovery from Anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 33 | 38
Participants | 7 | 3

3. Secondary Outcome: Delirium Rating Scale - Revised- 98 (DRS-R98) in Delirious Patients
Description: Measure Description: Delirium Rating Scale-Revised-98 (Severity items are rated on a scale of 0-3 and diagnostic items are rated on a scale of 0-2 or 0-3. The minimum score is 0. The maximum possible score for severity items is 39, while the maximum total score is 46. Higher scores indicate more severe delirium; score of 0 indicates no delirium.) Means and Standard Deviations were calculated from the maximum DRS-R98 score documented on Postoperative Day 1 and Day 2 for each participant who became delirious within each treatment arm.
Time Frame: Postoperative Day 1 and Day 2
Population: Participants With Delirium
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 3 | 2
score on a scale | 19.7 (8.0) | 19.0 (11.3)

ADVERSE EVENTS:
Time Frame: 30-day follow-up after surgery
Description: All adverse events (AE and SAE) were collected from the medical record and daily patient assessment using a customized instrument ("Health Questionnaire") which systematically probed for known side effects (fatigue, headache and next day somnolence).
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 3/41 | 0/39
Other Adverse Events (participants affected / at risk) | 13/41 | 13/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=41) | Placebo (N=39)
Bigeminy (Cardiac disorders) | 1 (1) | 0 (0) — Bigeminy noted during recovery from anesthesia
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Patient fell 5 days after original surgery
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) — Hypotension on POD #2 precluding discharge
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=41) | Placebo (N=39)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) — Facial Flushing
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fainting (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Reactive leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Sore throat (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Edema in limbs (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Eye disorders and eye pain (Eye disorders) | 2 (2) | 0 (0)
Foot pain (Surgical and medical procedures) | 1 (1) | 0 (0)
Hyperalertness (Nervous system disorders) | 0 (0) | 1 (1)
Restlessness (Nervous system disorders) | 0 (0) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Surgical procedure - other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT02324153/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT02324153/ICF_001.pdf